CLINICAL TRIAL: NCT01487096
Title: A Phase II Study of the Safety and Efficacy of Teriflunomide (HMR1726) in Multiple Sclerosis With Relapses
Brief Title: Safety and Efficacy of Teriflunomide (HMR1726) in Multiple Sclerosis With Relapses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMR1726D/2001
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — teriflunomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo (for teriflunomide),
  * two tablets once daily for 1 week then,
  * one tablet once daily for 35 weeks.
  Interventions: Drug: Placebo (placebo for teriflunomide)
- Teriflunomide 7 mg (Experimental): Teriflunomide 7 mg:
  * two tablets once daily for 1 week then,
  * one tablet once daily for 35 weeks.
  Interventions: Drug: Teriflunomide
- Teriflunomide 14 mg (Experimental): Teriflunomide 14 mg:
  * two tablets once daily for 1 week then,
  * one tablet once daily for 35 weeks.
  Interventions: Drug: Teriflunomide

INTERVENTIONS:
Drug: Teriflunomide — film-coated tablet
  oral administration
  Other Names: HMR1726
  Arms: Teriflunomide 14 mg; Teriflunomide 7 mg
Drug: Placebo (placebo for teriflunomide) — film-coated tablet
  oral administration
  Arms: Placebo

SUMMARY:
The primary objective of this study was to determine the safety and efficacy of teriflunomide in multiple sclerosis (MS) with relapses.

Secondary objectives were:

* To determine the effect of teriflunomide on additional magnetic resonance imaging (MRI) variables as well as clinical and quality of life measures.
* To investigate the pharmacokinetic and pharmacodynamic relationships.

DETAILED DESCRIPTION:
The total duration of the study period per participants was 46 weeks comprising 3 periods:

* a 4-week screening period,
* a 36-week double-blind treatment period,
* a 6-week post-treatment follow-up period.

Participants who successfully completed the double-blind treatment phase were offered the possibility to continue study treatment in the extension study LTS6048 - NCT00228163.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed multiple sclerosis [MS];
* Expanded Disability Status Scale [EDSS] score less or equal to 6;
* Two documented relapses in the previous 3 years, and one clinical relapse during the preceding year;
* Screening magnetic resonance imaging [MRI] scan fulfilling the criteria for a diagnosis of MS.

Exclusion Criteria:

* Clinically relevant cardiovascular, hepatic, hematologic, neurological, endocrine or other major systemic disease;
* Pregnant or nursing woman;
* Wish to parent children during the trial or following the trial (men and women were required to practice effective contraception during the trial and for 24 months after drug discontinuation);
* Prior treatment with interferon [IFN], gamma-globulin, glatiramer acetate, or other noncorticosteroid immunomodulatory therapies in the 4 months prior to the trial;
* Use of cladribine, mitoxantrone, or other immunosuppressant agents such as azathioprine, cyclophosphamide, cyclosporin, methotrexate or mycophenolate before enrollment;
* Any known condition or circumstance that would prevent in the investigator's opinion compliance or completion of the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2001-04; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
MRI assessment: number of unique active lesions per scan (T2/proton density and gadolinium-enhanced T1 scan analysis) | 36 weeks
  The number of unique active lesions per scan was calculated by dividing the sum of unique newly active lesions and unique persistently active lesions observed on treatment by the number of scans performed on treatment.
  Unique newly active lesions were all unique T1 and T2 lesions identified, one or more times, in a scan but not in the previous scan and, that had not been classified as unique newly active in any previous scan.
  Unique persistently active lesions were all unique T1 and T2 lesions identified, one or more times, in a scan and also in the previous scan.
Overview of Adverse Events [AE] | from first study drug intake up to 6 weeks after last intake or entry in the extension study, whichever came first
  AE are any unfavorable and unintended sign, symptom, syndrome, or illness observed by the investigator or reported by the participant during the study.

SECONDARY OUTCOMES:
MRI assessment: number of T1-enhancing lesions per scan | 36 weeks
  T1-enhancing lesions included:
  * Newly enhancing T1 lesions: lesions enhanced on the current T1 scan but not enhanced in any previous T1 scan.
  * Persistently enhancing T1 lesions: lesions enhanced on the current T1 scan and enhanced on the previous T1 scan.
MRI assessment: number of T2-lesions per scan | 36 weeks
  T2-lesions included:
  * New T2-lesions: lesions that appeared on the current T2 scan but were not visible on any previous T2 scans.
  * Newly enlarging T2-lesions: lesions that appeared enlarged on the current T2 scan but were stable on the previous T2 scan.
  * Persistently enlarging T2-lesions: further enlarged lesions on the current T2 scan categorized as new or enlarging on the previous T2 scan.
MRI assessment: Number of participants with no new lesions | 36 weeks
  New lesions included new T2 lesions, new enhanced T1 lesions and unique newly active lesions.
MRI assessment: Change from baseline in T2 burden of disease | 36 weeks
  T2 burden of disease was defined as the total volume of all T2 lesions.
Number of participants with progression on Expanded Disability Status Scale [EDSS] | 36 weeks
  EDSS is an ordinal scale in half-point increments that qualifies disability in patients with MS. It consists of 8 ordinal rating scales assessing seven functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation.
  EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS).
  Progression was defined as an increase in EDSS score by at least 1-point when baseline EDSS score ≤5.5 or an increase in EDSS score by at least 0.5-point in when baseline EDSS score >5.5.
Number of participants with MS relapse confirmed by Scripps Neurological Rating Scale [NRS] and EDSS scores. | 36 weeks
  A relapse was defined as the appearance, reappearance or worsening of a symptom attributable to MS. The change had to persist for at least 48 hours in the absence of fever and be preceded by stability or improvement for at least 30 days. Relapses were to be confirmed by Scripps NRS and EDSS scores.
  NRS is a scale that qualifies the degree of impairment from a neurological exam of the following systems: mentation and mood, cranial nerves, motor nerves, deep tendon reflexes, sensory nerves, cerebellum, gait/trunk/balance, bladder/bowel/sexual dysfunction.
  NRS score ranges from 0 to 100 (lower degree of impairment).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Director, Study Director — Clinical Science & Operation - sanofi-aventis
Locations (2):
- Canada, Toronto, Ontario, Canada
- sanofi-aventis France, Lyon, France

REFERENCES:
- [Result] O'Connor PW, Li D, Freedman MS, Bar-Or A, Rice GP, Confavreux C, Paty DW, Stewart JA, Scheyer R; Teriflunomide Multiple Sclerosis Trial Group; University of British Columbia MS/MRI Research Group. A Phase II study of the safety and efficacy of teriflunomide in multiple sclerosis with relapses. Neurology. 2006 Mar 28;66(6):894-900. doi: 10.1212/01.wnl.0000203121.04509.31. PMID 16567708
- [Derived] Comi G, Freedman MS, Meca-Lallana JE, Vermersch P, Kim BJ, Parajeles A, Edwards KR, Gold R, Korideck H, Chavin J, Poole EM, Coyle PK. Prior treatment status: impact on the efficacy and safety of teriflunomide in multiple sclerosis. BMC Neurol. 2020 Oct 6;20(1):364. doi: 10.1186/s12883-020-01937-4. PMID 33023488